CLINICAL TRIAL: NCT01736397
Title: A Phase 2 Study of KRX-0502 (Ferric Citrate) in Managing Serum Phosphorus and Iron Deficiency in Anemic Subjects With Stage III to V Chronic Kidney Disease Not on Dialysis
Brief Title: Ferric Citrate in Managing Serum Phosphorus and Iron Deficiency in Anemic Chronic Kidney Disease (CKD) Subjects Not on Dialysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KRX-0502-204
Record Dates: First submitted 2012-11-16; First posted 2012-11-29 (Estimated); Results first posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Iron Deficiency; Iron Deficiency Anemia
Keywords: CKD; Chronic Kidney Disease; Phosphorus; Iron Deficiency; Iron Deficiency Anemia; Elevated Phosphorus
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency; Renal Insufficiency, Chronic | interventions — ferric citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric Citrate (Experimental): Ferric citrate will be taken with or within one hour of meals or snacks. The starting dose of ferric citrate is 3 tablets/day and titrated by the subject's serum phosphorus results at each treatment visit.
  Interventions: Drug: Ferric Citrate
- Placebo (Placebo Comparator): Placebo will be taken with or within one hour of meals or snacks. The starting dose of placebo is 3 tablets per day and titrated by the subject's serum phosphorus results at each treatment visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric Citrate — Dose depends on serum phosphorus levels collected at each study visit.
  Other Names: KRX-0502
  Arms: Ferric Citrate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if KRX-0502 (ferric citrate) is a safe and effective treatment for the management of serum phosphorus levels and iron deficiency in anemic chronic kidney disease (CKD) stage 3-5 subjects not on dialysis. Total length of treatment is approximately 12 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, three-period, multi-center clinical trial. Following a Screening and Qualification Period and a two-week Washout Period (for those subjects entering the study on a phosphate binder), eligible subjects will be randomized in a 1:1 ratio to receive either KRX-0502 (ferric citrate) or placebo for up to approximately 12 weeks. The purpose of this study is to determine if KRX-0502 (ferric citrate) is a safe and effective treatment for the management of serum phosphorus levels and iron deficiency in anemic CKD subjects not on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Stage III to V Chronic Kidney Disease
* Serum Phosphorus 4.0-6.0 mg/dL prior to Randomization
* Ferritin 300 ng/mL or less
* Transferrin Saturation (TSAT) 30% or less
* Hemoglobin >9.0 and <12.0 g/dL
* Must consume a minimum of 2 meals per day

Exclusion Criteria:

* Parathyroidectomy within 24 weeks of study
* gastrointestinal bleed or inflammatory bowel disease within 12 weeks of study
* Requirement for dialysis or kidney injury within 8 weeks of study
* Absolute requirement for oral iron, intravenous iron, Erythropoiesis-Stimulating Agent, blood transfusions, and Sensipar during the study
* Absolute requirement for calcium-, magnesium-, or aluminum-containing drugs with meals
* Absolute requirement for vitamin C, niacin, or nicotinamide outside of multivitamins
* History of hemochromatosis
* Allergy to iron products
* History of malignancy in last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Block, MD, Study Chair; Glenn Chertow, MD, Study Chair; Steven Fishbane, MD, Study Chair
Locations (20):
- United States (20):
  - Tempe, Arizona
  - La Mesa, California
  - Sacramento, California
  - Denver, Colorado
  - Edgewater, Florida
  - Miami, Florida
  - Meridian, Idaho
  - Evergreen Park, Illinois
  - Bethesda, Maryland
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Pontiac, Michigan
  - Reno, Nevada
  - Great Neck, New York
  - Mineola, New York
  - Asheville, North Carolina
  - Wilmington, North Carolina
  - Orangeburg, South Carolina
  - Houston, Texas
  - San Antonio, Texas

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Block GA, Fishbane S, Rodriguez M, Smits G, Shemesh S, Pergola PE, Wolf M, Chertow GM. A 12-week, double-blind, placebo-controlled trial of ferric citrate for the treatment of iron deficiency anemia and reduction of serum phosphate in patients with CKD Stages 3-5. Am J Kidney Dis. 2015 May;65(5):728-36. doi: 10.1053/j.ajkd.2014.10.014. Epub 2014 Nov 4. PMID 25468387

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferric Citrate: Ferric citrate will be taken with or within one hour of meals or snacks. The dose of ferric citrate will depend on the patient's serum phosphorus results at each treatment visit.
  Ferric Citrate: Dose depends on serum phosphorus levels collected at each study visit.
- Placebo: Placebo will be taken with or within one hour of meals or snacks. The number of placebo pills will depend on the patient's serum phosphorus results at each treatment visit.
  Placebo
Period: Overall Study
Arm/Group | Ferric Citrate | Placebo
Started | 75 | 74
Completed | 61 | 50
Not Completed | 14 | 24
Not completed — Lack of Efficacy | 1 | 11
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 6 | 3
Not completed — Not stated | 1 | 4

BASELINE CHARACTERISTICS:
Population: One subject on placebo was randomized but never received drug and so was excluded from the safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Citrate | Placebo | Total
Number analyzed (Participants) | 75 | 73 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 34 | 65
  >=65 years | 44 | 39 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (12.15) | 64.5 (13.55) | 65.1 (12.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 45 | 96
  Male | 24 | 28 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 21 | 36
  Not Hispanic or Latino | 60 | 52 | 112
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 16 | 32
  White | 59 | 56 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75 | 73 | 148
Chronic kidney disease (CKD), stage at baseline [Count of Participants; unit: Participants] — The stage of CKD disease was measured by the estimated glomerular filtration rate (eGFR), where CKD Stage III relates to better kidney function compare to CKD Stage V, that has worse kidney function.
  Stage III: eGFR 30-59 mL/min/1.73 m2 Stage IV eGFR 15-29 mL/min/1.73 m2 Stage V eGFR<15 mL/min/1.73 m2 Other eGFR >=60 mL/min/1.73 m2
  Participants
    Stage III | 14 | 16 | 30
    Stage IV | 39 | 39 | 78
    Stage V | 21 | 17 | 38
    Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Transferrin Saturation (TSAT) From Baseline to End of Treatment
Description: The difference in TSAT between the value at the end of treatment (week 12) minus the baseline measurement.
Time Frame: 12 Weeks
Population: Efficacy analyses were based on Intent-to-Treat (ITT) population, which consisted of all randomized subjects who had a baseline laboratory value, had taken at least 1 dose of study drug, & had at least 1 post-baseline laboratory value. ANCOVA with Last observation carried forward (LOCF) methodology was used.
Measure: Mean (Standard Deviation); unit: % saturation
Arm/Group | Ferric Citrate | Placebo
Number analyzed (Participants) | 72 | 69
% saturation
  Baseline | 21.6 (7.44) | 21.0 (8.26)
  Week 12 | 31.7 (14.19) | 20.0 (7.55)

2. Primary Outcome: Change in Serum Phosphorus Levels From Baseline to End of Treatment
Description: The difference in serum phosphorus between the value at the end of treatment (week 12) minus the baseline measurement.
Time Frame: 12 Weeks
Population: The efficacy analyses were based on the ITT population. The Intent-to-Treat (ITT) population consisted of all subjects who were randomized into the study, had a baseline laboratory value, had taken at least 1 dose of study drug, and had at least 1 post-baseline laboratory value. ANCOVA with LOCF methodology was used.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ferric Citrate | Placebo
Number analyzed (Participants) | 72 | 69
mg/dL
  Baseline | 4.5 (0.61) | 4.7 (0.60)
  12 weeks | 3.9 (0.58) | 4.4 (0.75)

3. Secondary Outcome: Change in Ferritin Levels From Baseline to End of Treatment
Description: The difference in ferritin levels between the value at the end of treatment (week 12) minus the baseline measurement.
Time Frame: 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ferric Citrate | Placebo
Number analyzed (Participants) | 72 | 69
ng/mL
  Baseline | 115.8 (83.11) | 110.0 (80.88)
  Week 12 | 189.4 (122.16) | 105.6 (93.87)

4. Secondary Outcome: Change in Hemoglobin Levels From Baseline to End of Treatment
Description: The difference in hemoglobin levels between the value at the end of treatment (week 12) minus the baseline measurement.
Time Frame: 12 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferric Citrate | Placebo
Number analyzed (Participants) | 72 | 69
g/dL
  Baseline | 10.5 (0.81) | 10.6 (1.07)
  Week 12 | 11.0 (1.03) | 10.4 (1.14)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: One subject on placebo was randomized but never received drug and so was excluded from the safety population
Arm/Group | Ferric Citrate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 2/73
Serious Adverse Events (participants affected / at risk) | 6/75 | 9/73
Other Adverse Events (participants affected / at risk) | 52/75 | 43/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Citrate (N=75) | Placebo (N=73)
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Congestive Cardiac Failure (Cardiac disorders) | 1 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Renal Failure Chronic (Renal and urinary disorders) | 0 | 1
COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Accelerated Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Citrate (N=75) | Placebo (N=73)
Faeces Discolored (Gastrointestinal disorders) | 24 | 0
Diarrhoea (Gastrointestinal disorders) | 15 | 4
Constipation (Gastrointestinal disorders) | 14 | 4
Nausea (Gastrointestinal disorders) | 5 | 5
Vomiting (Gastrointestinal disorders) | 4 | 4
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 4
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 2 | 1
Oedema (General disorders) | 2 | 1
Oedema Peripheral (General disorders) | 3 | 1
Foot Fracture (Injury, poisoning and procedural complications) | 2 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days